CLINICAL TRIAL: NCT04585438
Title: Evaluation of Trans-mucosal Bio-adhesive Discs of Diclofenac Potassium on the Anesthetic Success and Postoperative Pain in Patients With Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Yousef Soliman, Ahmed Yousef Soliman, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO:3-5-5
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Irreversible Pulpitis; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Diclofenac

STUDY DESIGN:
Intervention Model Description: Trial Design: Randomized Clinical Trial (Parallel Group) Two Arms Allocation Ratio: 1:1 Framework: Superiority
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Allocation sequence generation: The co-supervisor who will assign the participants to either groups and will be the only one to know whether A or B represents the intervention or the control group. The principal investigator will enroll according to the previously mentioned eligibility criteria. The participant will drag an envelope and will be given a number. The patient will be allocated to either intervention or control group after contacting the co-supervisor to reveal the assigned group of the current patient according to the generated random sequence. The patient and the operator will not know the intervention done. The treatment groups will remain anonymous at the end of the study during assessment by the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single trans-mucosal bio-adhesive disc containing Diclofenac Potassium (Experimental): Premedication 1 hour before starting endodontic treatment.
  Interventions: Drug: Diclofenac Potassium
- Placebo Control (Placebo Comparator): Premedication 1 hour before starting endodontic treatment. Identically-appearing trans-mucosal bio-adhesive disc (Does not contain medication)
  Interventions: Drug: Diclofenac Potassium

INTERVENTIONS:
Drug: Diclofenac Potassium — The drug will be used as a transparent disc applied to the mucosa
  Other Names: Cataflam

SUMMARY:
The aim of the proposed study is to compare the effect of single dose of Diclofenac Potassium premedication as trans-mucosal bio-adhesive discs versus placebo on the effectiveness of the inferior alveolar nerve block and postoperative pain in patients with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
One of the challenging goals of root canal therapy is to relieve the pain associated with irreversible pulp inflammation. Pain control especially in the early stages of treatment, is critical and can enhance the confidence of both the patient and the dentist. Irreversible pulpitis pain is sometimes difficult to be managed through the use of local anesthetics solely. Inadequate pain control during treatment may contribute to the development of peripheral and central sensitization leading to greater pain during recovery. Various mechanisms have been proposed to explain the failure of local anesthetics including anatomic variations such as; cross innervations and accessory innervations, tachyphylaxis of anesthetic solutions, and activation of nociceptors including tetrodotoxin (TTX).Strategies to control intra-operative endodontic pain include preoperative administration of analgesics, supplemental infiltrations, the use of different local anesthetic solutions, intra-osseous and periodontal injections, a repeat inferior alveolar nerve block. Prescribing drugs prior to treatment may enhance the patient's attitude and reduce the apprehension during endodontic therapy. Non-steroidal anti-inflammatory drugs (NSAIDs) are the most common category of medications recommended for pain relief. They act by inhibition of prostaglandin synthesis by inhibition of cyclooxygenase pathway. Although, pulpectomy and removal of the inflamed pulpal tissues eliminates endodontic pain, post-operative pain and discomfort are common side effects. Many patients may still experience mild to extreme pain even after therapy. Diclofenac has shown a substantial reduction of post-endodontic pain when administered preoperatively in a single oral dose since it holds anti-inflammatory, antipyretic and analgesic effects. It acts primarily by inhibition of COX 1 and COX 2, thus inhibiting the prostaglandin synthesis. COX 1 is expressed throughout the body and has a role in protection of stomach mucosa, kidney function and platelet action. Numerous studies have clearly documented that the risk of upper gastrointestinal complications increases with increasing doses as well as increasing frequency of use. Additionally, when taken through oral route, only 50% of the absorbed dose of Diclofenac becomes available systematically, due to its first pass metabolism. Trans-mucosal drug delivery offers distinct advantages over oral administration such as avoiding hepatic first-pass metabolism, less dosing frequency, improved patient compliance, reduction in fluctuation in steady-state levels. In addition, there is a reduced intensity of local or systemic side effects, increased safety margin and maximum utilization of drug and reduction in the total amount of drug administered while achieving target delivery in odontogenic region.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are free from any physical or mental handicapping condition with no underlying systemic disease.
* Age between 18-50 years old.
* Males & Females.
* Mandibular permanent molar teeth with:

  * Preoperative sharp pain.
  * Positive response of pulp tissue to cold pulp tester (ethyl chloride spray ) and electric pulp tester
  * Normal periapical radiographic appearance or slight widening in lamina dura using periapical index (PAI) score 1 as normal periapical structures or 2 as small changes in bone structures.
  * Patients' acceptance to participate in the trial.
  * Patients who can understand pain scale and can sign the informed consent

Exclusion Criteria:

* Medically compromised patients: Pain levels and healing following treatment would be compromised as these patients have shown higher incidence of pain and lower healing rate.
* Pregnant women: Avoid radiation exposure, anesthesia, and medication.
* If analgesics have been administrated by the patient during the past 24 hours preoperatively might alter their pain perception.
* Patients reporting bruxism or clenching: Avoid further pressure on an already inflamed tooth inducing subsequent irritation and inflammation.
* Teeth with necrotic pulp, acute periapical abscess and swelling: Need special treatment steps, it could influence initiation and progression of postoperative pain.
* Greater than grade I mobility or pocket depth greater than 5mm. Need special surgical and/or periodontal therapy.
* No restorability: Hopeless tooth.
* Immature teeth.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09-21 (Estimated); Primary Completion 2022-09-21 (Estimated); Study Completion 2022-09-22 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the inferior alveolar nerve block during cold test or any stage of access cavity preparation or instrumentation in patients with irreversible pulpitis. | During endodontic treatment
  the outcome will be measured with Heft-parker visual analogue scale (VAS) in which no or mild pain (Heft-Parker VAS rating less than 54mm) will be considered as anesthetic success and moderate or severe pain (Heft-parker VAS rating greater than 54mm) will be considered as anesthetic failure.

SECONDARY OUTCOMES:
Intensity of postoperative pain | at 6, 12, 24, 48 hours after the end of endodontic treatment.
  the outcome will be measured using Heft-parker VAS